CLINICAL TRIAL: NCT04975152
Title: Neoadjuvant Cemiplimab in Newly Diagnosed or Recurrent Stage I-II Merkel Cell Carcinoma and Locoregionally Advanced Cutaneous Squamous Cell Carcinoma: Safety and Biomarker Analysis
Brief Title: Neoadjuvant Cemiplimab in Newly Diagnosed or Recurrent Stage I-II Merkel Cell Carcinoma and Locoregionally Advanced Cutaneous Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20794
Record Dates: First submitted 2021-07-22; First posted 2021-07-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Merkel Cell Carcinoma; Cutaneous Squamous Cell Carcinoma
Keywords: Skin Cancer
MeSH Terms: conditions — Carcinoma, Merkel Cell; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant Cemiplimab Treatment (Experimental): Participants will receive cemiplimab 350 mg IV at least 3 weeks prior to surgical resection. After surgery they will continue to receive 350 mg cemiplimab every 3 weeks for up to 8 additional doses.
  Interventions: Drug: Cemiplimab-Rwlc

INTERVENTIONS:
Drug: Cemiplimab-Rwlc — Flat dose of cemiplimab-rwlc 350 mg IV every 3 weeks, up to 9 cycles.
  Other Names: Libtayo

SUMMARY:
The goal of this clinical research study is to determine if Cemiplimab-rwlc (called Cemiplimab in this document) given prior to tumor resection surgery is safe and effective in treating (1) Merkel Cell Carcinoma or (2) Cutaneous Squamous Cell Carcinoma (CSCC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of Merkel cell carcinoma (MCC).
* Clinical stage I-II MCC (AJCC 8th edition) either newly diagnosed or previously diagnosed with recent disease recurrence. This includes patients with a previous diagnosis of clinical Stage I-II who present with local or regional disease recurrence.
* Patients must be considered candidates for wide local surgical excision and may be candidates for sentinel lymph node biopsy. If sentinel biopsy is determined to not be clinically indicated then it would not be required to be completed and only the tumor excision would be required.
* Patients with stage III to stage IV (M0) CSCC of the head/neck, extremity, or trunk, and selected patients with stage II CSCC (≥3 cm longest diameter lesion in an aesthetically-sensitive region), for whom surgery is planned.
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged at least 18 years
* ECOG performance Status of 0, 1, or 2
* Adequate baseline laboratory assessments within 28 days of study registration:

  1. Adequate hepatic function: i. Total bilirubin ≤1.5 x upper limit of normal (ULN) (NOTE: For patients with Gilbert's syndrome, total bilirubin ≤3 x ULN) ii. Transaminases (aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) ≤3 x ULN iii. Alkaline phosphatase (ALP) ≤2.5 x ULN
  2. Adequate renal function: Serum creatinine ≤1.5 x ULN or estimated creatinine clearance (CrCl) >30 mL/min according to the method of Cockcroft and Gault.
  3. Adequate bone marrow function: i. Hemoglobin ≥9.0 g/dL ii. Absolute neutrophil count (ANC) ≥1.0 x 109/L iii. Platelet count ≥75 x 109/L
* Patients who are HIV+ with undetectable HIV viral load are eligible.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 months after the end of cemiplimab administration.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner

Exclusion Criteria:

* Concurrent malignancy other than localized CSCC and/or history of malignancy other than Merkel cell carcinoma within 3 years of date of registration on the study, except for tumors with negligible risk of metastasis or death, such as adequately treated (BCC) of the skin, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast, or low- risk early stage prostate adenocarcinoma (T1-T2aN0M0 and Gleason score ≤6 and prostate-specific antigen (PSA) ≤10 ng/mL) for which the management plan is active surveillance, or prostate adenocarcinoma with biochemical-only recurrence with documented PSA doubling time of >12 months for which the management plan is active surveillance.
* Patients with hematologic malignancies (eg, chronic lymphocytic leukemia [CLL]).
* Ongoing or recent (within 5 years of registration date) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-related adverse events (irAEs). Further, patients requiring chronic immune-suppressive therapy are excluded. The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment.
* Pregnancy or lactation.
* Has participated in a study of an investigational agent or an investigational device within weeks of the enrollment date.
* Receipt of a live vaccine within 28 days of the registration date.
* Has had prior systemic anti-cancer immunotherapy for MCC. Examples of immune modulating agents include but are not limited to blockers of CTLA-4, 4-1BB (CD137), or OX-40, therapeutic vaccines, anti-PD-1/PD-L1.
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of cemiplimab/placebo.

NOTE: Patients who require brief course of corticosteroids (eg, prophylaxis for imaging assessments due to hypersensitivity to contrast agents) are not excluded. People taking steroids for physiologic replacement (ie, adrenal insufficiency) are NOT excluded.

- Has received treatment with an approved anticancer systemic therapy within 4 weeks of the registration date or has not yet recovered (ie, ≤ grade 1 or baseline) from any acute toxicities except for laboratory changes as described in the inclusion criteria.

NOTE: Patients receiving bisphosphonates or denosumab are not excluded.

* Prior allogeneic stem cell transplantation, or autologous stem cell transplantation.
* Patients who have permanently discontinued anti-cancer immune modulating therapies due to drug-related toxicity.
* Encephalitis, meningitis, or uncontrolled seizures in the year prior to screening.
* Patients with myocardial infarction within 6 months prior to the registration date.
* Any infection requiring hospitalization and/or intravenous antibiotic therapy within 2 weeks of the registration date.
* Active tuberculosis.
* Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus (HBV or HCV) infection; or diagnosis of immunodeficiency.

NOTES:

* Patients with known HIV infection who have controlled infection (undetectable viral load (HIV RNA PCR) and CD4 count above 350, either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
* Patients with HBV (hepatitis B surface antigen positive; HepBsAg+) who have controlled infection (serum HBV DNA PCR that is below the limit of detection AND receiving anti- viral therapy for HBV) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug.

Patients who are HCV antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by PCR, either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.

* History of immune related pneumonitis within the last 5 years.
* History of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in the radiation field is permitted as long as pneumonitis resolved ≥6 months prior to the registration date.
* History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments.
* Known hypersensitivity or allergy to any of the excipients in the cemiplimab drug product.
* Patients with a history of solid organ transplant (exception: patients with prior corneal transplant are not excluded).
* Any medical co-morbidity, physical examination finding, or metabolic dysfunction, or clinical laboratory abnormality that, in the opinion of the investigator, renders the patient unsuitable for participation in a clinical trial due to high safety risks and/or potential to affect interpretation of results of the study.
* Known psychiatric or substance abuse disorders that would interfere with participation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events Related to Study Treatment | Beginning of treatment to end of follow up, up to 3 years
  Number of participants with adverse events after receiving at least one dose of cemiplimab

SECONDARY OUTCOMES:
Relapse Free Survival | Up to 3 years
  Relapse Free Survival (RFS) is defined as the time from study enrollment until disease recurrence or death.
Overall Survival | Up to 3 years
  Overall Survival (OS) is defined as the time from study enrollment until death.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided